CLINICAL TRIAL: NCT07074665
Title: A Phase II Randomised Trial to Evaluate the Safety and Immunogenicity of a R21/Matrix-M Booster Vaccine at Two Different Doses in Burkinabe School Children
Brief Title: Dose Finding Trial of R21/Matrix-M in School Children
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAC101
Record Dates: First submitted 2025-06-23; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Malaria (Plasmodium Falciparum)
Keywords: Malaria Vaccine; R21/Matrix-M
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Participants in this arm will be given one dose of 5µg R21/50µg Matrix-M
  Interventions: Biological: 5µg R21/50µg Matrix-M
- Group B (Experimental): Participants in this arm will be given one dose of 10µg R21/50µg Matrix-M
  Interventions: Biological: 10µg R21/50µg Matrix-M

INTERVENTIONS:
Biological: 5µg R21/50µg Matrix-M — R21/Matrix-M is a vaccine against P. falciparum malaria, which has WHO prequalification and policy recommendation in children over 5 months old in malaria endemic areas. The standard paediatric dose is 5µg R21/50µg Matrix-M.
  Arms: Group A
Biological: 10µg R21/50µg Matrix-M — R21/Matrix-M is a vaccine against P. falciparum malaria, which has WHO prequalification and policy recommendation in children over 5 months old in malaria endemic areas. 10µg R21/50µg Matrix-M is the standard adult dose.
  Arms: Group B

SUMMARY:
This trial is a double-blind, randomised, trial recruiting participants from the R21 phase IIb trial (VAC 076) which took place between May 2019 and July 2023 in Nanoro, Burkina Faso.

Participants (n=30-40) who have previously received four doses of the 5µg R21/50µg Matrix-M malaria vaccine in VAC 076 will be randomised to receive either 5µg R21/50µg Matrix-M or 10µg R21/50µg Matrix-M. Safety and immunogenicity of a booster at school age at these two different doses will be assessed. Participants will be followed up for one year after the booster.

ELIGIBILITY:
Inclusion Criteria:

* The child received four doses of R21/Matrix-M in the phase IIb study evaluating R21/MatrixM in Nanoro, Burkina Faso (VAC 076).
* Signed informed consent/thumb-printed and witnessed informed consent obtained from the parent(s)/guardian(s) of the child to join the trial.
* The investigator believes that the parents/guardians can and will comply with the requirements of the protocol if the child is enrolled in the study.
* The child is a permanent resident of the study area and is expected to remain a resident for the duration of the trial.

Exclusion Criteria:

* The child is enrolled in another malaria vaccine trial.
* The child has a history of allergic disease or reactions likely to be exacerbated by any component of the malaria vaccine.
* The child has a history of allergic reactions, significant IgE-mediated events or anaphylaxis to previous immunisations.
* The child has major congenital defects.
* The child has anaemia associated with clinical signs of symptoms of decompensation, or a haemoglobin of ≤ 5.0 g/dL.
* The child has been administered immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
* The child has malnutrition requiring hospital admission.
* The child has an acute or chronic, clinically significant pulmonary, cardiovascular, gastrointestinal, endocrine, neurological, skin, hepatic or renal functional abnormality, as determined by medical history, physical examination or laboratory tests.
* Children currently meeting the WHO criteria for HIV disease of stage 3 or 4 severity. A previous history of stage 3 or 4 disease is not an exclusion. Note: There will be no routine testing for HIV. Positive diagnoses will be recorded at screening if known.
* The child has received an investigational drug or investigational vaccine other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* The child is currently participating in another clinical trial if likely to affect data interpretation of this trial.
* The child has any significant disease, disorder or situation which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Reactogenicity | 7 days after vaccination
  Reactogenicity of an additional late booster of R21/Matrix-M at different doses, in school age children living in Burkina Faso. This will be measured through: 1) the occurrence of solicited local reactogenicity signs and symptoms for 7 days following the vaccination and 2) the occurrence of solicited systemic reactogenicity signs and symptoms for 7 days following the vaccination.
Safety - unsolicited AEs | 28 days following vaccination
  Safety of an additional late booster of R21/Matrix-M at different doses, in school age children living in Burkina Faso will be assessed through the occurrence of unsolicited adverse events for 28 days following the vaccination.

SECONDARY OUTCOMES:
Immunogenicity | At baseline and one, six and twelve months after vaccination
  Humoral immunogenicity by anti-CSP antibody concentrations after school age booster of R21/Matrix-M at different doses.
Safety - SAEs | 1 year after vaccination
  Serious adverse events (SAEs) following school age booster vaccination.
Safety - deaths | 1 year after vaccination
  Any deaths following school age booster vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Unité de Recherche Clinique de Nanoro (URCN), Nanoro, Burkina Faso

IPD SHARING:
Plan to Share IPD: Yes
Yes de-identified individual participant data collected in this study may be made available to other researchers outside the main trial team. This could include data on vaccinations, health, demographics or immunology results. Any proposals for using the study data will be reviewed and approved by the sponsor trial team.